CLINICAL TRIAL: NCT01361269
Title: Multicentre Evaluation of Fosmidomycin and Clindamycin in the Treatment of Acute Uncomplicated Plasmodium Falciparum Malaria in African Children
Brief Title: Evaluation of Fosmidomycin and Clindamycin in the Treatment of Acute Uncomplicated Plasmodium Falciparum Malaria
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zentopharm GmbH (Industry)
Collaborators: Albert Schweitzer Hospital (Other); Centro de Investigacao em Saude de Manhica (Other)
Responsible Party: Saadou Issifou, Medical Research Unit, Albert Schweitzer Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FosClinChildren
Record Dates: First submitted 2011-05-24; First posted 2011-05-26 (Estimated); Last update posted 2011-05-26 (Estimated); Status verified 2011-05

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria | interventions — fosmidomycin; Clindamycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fosmidomycin and clindamycin treatment (Experimental): All the subject will be given fosmidomycin 30mg/kg/dose + clindamycin 10mg/kg/dose twice daily for three days (total daily dose fosmidomycin 60mg/kg, clindamycin 20mg/kg).
  Interventions: Drug: Fosmidomycin and clindamycin

INTERVENTIONS:
Drug: Fosmidomycin and clindamycin — The study drugs will be co-administered under supervision by a study physician or nurse in doses of fosmidomycin 30mg/kg/dose + clindamycin 10mg/kg/dose twice daily for three days (total daily dose fosmidomycin 60mg/kg, clindamycin 20mg/kg).

SUMMARY:
Few efficient drugs for malaria treatment are available so far. Due to increased exposure of these drugs and due to the high risk of development of drug resistant strains of Plasmodium falciparum, new drug combinations have to be actively investigated. The investigators will test the efficiency, safety and tolerance of combined fosmidomycin and clindamycin treatment in acute uncomplicated malaria in children aged 3-10 years.

DETAILED DESCRIPTION:
Few efficient drugs for malaria treatment are available so far. Due to increased exposure of these drugs and due to the high risk of development of drug resistant strains of Plasmodium falciparum, new drug combinations have to be actively investigated. The goal of this study is to assess a new drug combination, fosmidomycin-clindamycin. The primary objective of the study is to assess and compare the efficacy, safety and tolerance (between sites) of fosmidomycin and clindamycin when co-administered orally over three days in the treatment of acute uncomplicated Plasmodium falciparum malaria in children in Mozambique and Gabon.

The secondary objective is to differentiate between recrudescent parasitaemia and reinfection in the event of recurrent parasitaemia developing within the 28-day follow-up period, to determine the population pharmacokinetics of fosmidomycin when co-administered orally with clindamycin and to compare the in vitro sensitivity of isolates of Plasmodium falciparum to fosmidomycin.

The trial will include 100 children aged 3-10 years, divided between clinical sites of Gabon and Mozambique.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged three to ten years
* Body weight ≥12kg
* Acute (symptoms lasting less than 14 days) uncomplicated P falciparum malaria
* Asexual parasitaemia between 1,000/µL and 200,000/µL
* Ability to tolerate oral therapy
* Willingness of the parent or guardian to provide informed signed consent

Exclusion Criteria:

* Symptoms/signs of severe malaria, according to WHO criteria (see appendix I)
* Body weight <12kg
* Other concomitant plasmodial infections (P vivax, P ovale, P malariae)
* Severe malnutrition with weight for height <70% (according to WHO tables) or clinical kwashiorkor
* Gastro-intestinal disturbance with persistent vomiting (> three episodes within previous 24 hours) and/or diarrhoea (> 5 loose stools in the preceding 24 hours)
* Concomitant disease masking assessment of response including sickle cell disease and severe cardiac, hepatic or renal impairment
* Packed cell volume (PCV) on arrival <22%
* Adequate anti-malarial treatment within previous 7 days
* Inability to tolerate oral therapy
* Parent or guardian deemed to be unsupportive
* On co-trimoxazole prophylaxis
* Any known allergies to the investigational products

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2011-06; Primary Completion 2011-09 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Cure rate | Day 28
  Cure rate at day 28 will be determined by PCR

SECONDARY OUTCOMES:
cure rate | day 7
  The secondary endpoints will be the cure rate on Day 7 and the parasite and fever clearance times.

CONTACTS AND LOCATIONS:
Overall Officials: Saadou Issifou, MD PhD, Principal Investigator — Medical Research Unit, Albert Schweitzer Hospital
Locations (1):
- Medical Research Unit, Albert Schweitzer Hospital, Lambaréné, Gabon